CLINICAL TRIAL: NCT02969434
Title: Accuracy of the Brief Pain Inventory in Identifying Sleep Disturbances in Chronic Pain Patients
Brief Title: Chronic Pain and Assessment of Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1/027/16
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep questionnaires assessment tools (Experimental): Interventions are 3 tools to assess sleep: Verran Snyder Halpern sleep scale, the Pain and Sleep Questionnaire 3 Item Index (PSQ-3) and the Pittsburg Sleep Quality Index (PSQI).
  Interventions: Other: Sleep assessment tools

INTERVENTIONS:
Other: Sleep assessment tools — Interventions are 3 tools to assess sleep: Verran Snyder Halpern sleep scale, the Pain and Sleep Questionnaire 3 Item Index (PSQ-3) and the Pittsburg Sleep Quality Index (PSQI).

SUMMARY:
Sleep impairments reliably predict worsened chronic pain and correlate with visual analogue pain scores. Therapies targeted at improving sleep, including cognitive behavioral therapy, improve both sleep quality and also pain management, and reduce interference of pain with daily activities. As effective pain relief decreases sleep disturbances, improvement in sleep has been proposed as marker of effective pain management. Hence it is useful to evaluate sleep disturbances in chronic pain population both in clinical and research setting. There are many tools to evaluate sleep quality; the routinely used simple brief pain inventory (BPI) has a single question about sleep. We will compare three dedicated sleep measures to the BPI in patients with chronic pain.

DETAILED DESCRIPTION:
The prevalence of sleep disturbances including insomnia is high in chronic pain patients and is known to contribute to the maintenance of chronic pain. A large survey estimated that chronic pain of moderate to severe intensity occurs in 19% of adult Europeans, and that 50% of this cohort reported feeling tired all the time. Studies using specific sleep assessment tools have found that up to 50% of patients complain of poor sleep and 40% have clinically defined insomnia.

Though association between sleep and pain is well established, it is still unclear about the direction of causality. A recent narrative review has found that sleep impairments reliably predict worsening of chronic pain and correlate with higher visual analogue pain scores. Therapies targeted at improving sleep hygiene, including cognitive behavioral therapy, have been shown to not only improve sleep quality, but also pain management and reduce the degree to which pain interfered with daily activities. As effective pain relief decreases sleep disturbances, improvement in sleep has been proposed as marker of effective pain management.8 Hence it is useful to evaluate sleep disturbances in chronic pain population both in clinical and research setting.

There are at least 30 different sleep evaluation scales and questionnaires. Previous works have used several different tools to quantify the prevalence and severity of sleep disturbance in chronic pain patients. The most commonly used tools are the Pittsburgh Sleep Quality Index (PSQI) and the Medical Outcomes Study (MOS) Sleep Scale. The PSQI has an extensive body of evidence in detecting primary insomnia, demonstrating a high test-retest reliability and contains domains which are of importance when measuring sleep disturbance in chronic pain. However, none of the aforementioned tools directly assesses the impact of pain on sleep, and are as such not capable of establishing a direct link between sleep disturbance and chronic pain. Chronic Pain Sleep Inventory (CPSI) and Pain and Sleep Questionnaires (PSQ) were developed to assess the impact of pain on pain related sleep disturbances. These multidimensional items were abbreviated to Sleep Pain Index (SPI) and Pain and Sleep three-item index (PSQ-3) and specifically targeted at assessing sleep disturbance in patients with chronic pain. Both SPI and PSQ- 3 have been tested for their reliability and validity. The Verran Snyder-Halpern (VSH) scale uses visual analogue scales to describe sleep quality, latency and disturbance but none of these questionnaires have been widely adopted either in research setting or clinical practice. Though the reasons are not known, people may find multi-items dedicated questionnaires as cumbersome and overwhelming. One way to circumvent the issue is to utilize a single item questionnaire or even use a single item on the widely used pain questionnaire. Single item numerical rating scales to measure sleep quality have shown modest correlation with the MOS sleep scale and may be of particular benefit when repeated measurements are used due to their simple nature.

Brief Pain Inventory (BPI) is one of the most widely used measurement tool and is advocated as one of the core outcomes tool for pain clinical trials. BPI provides an overall picture of pain status and its interference with general health and serves to help monitor response to treatment with time. Included in the BPI is a single numerically rated score assessing the degree to which pain interferes with sleep. This item has the potential to detect the impact of pain on pain related sleep disturbances thereby insomnia and therefore lead to treatment. Validation of this commonly used questionnaire BPI, against a formal sleep assessment tools would not only allow identification of patients with significant sleep disturbance and facilitate prompt targeted treatment but also help to evaluate the pain treatment.

ELIGIBILITY:
Inclusion Criteria:

Aged 16 or over Chronic pain Fluent in English Able to report on their health and pain status (neurologically stable)

Exclusion Criteria:

Under 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Recruitment of 50 patients | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Saravanakumar F Kanakarajan, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen/NHS Grampian, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No